CLINICAL TRIAL: NCT05746247
Title: Improving Diagnosis and Clinical Management of Familial Hypercholesterolemia Through Integrated Machine Learning, Implementation Science, and Behavioral Economics
Acronym: BEAT FH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Family Heart Foundation (Unknown); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 849516
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Familial Hypercholesterolemia
Keywords: machine learning; FIND FH
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: For the pilots, for patients with a PCP within the healthcare system, we are testing 2 different centralized referral models to increase the # of patients that see a lipid specialist (active choice vs default).
  For patients without a PCP within the health system, we are testing out health system mediated outreach vs Family Heart Foundation mediated outreach in order to increase the number of patients who make an appointment with a lipid specialist.
  For Phase 3: There will be 2 arms. Arm 1) Penn PCP: For patients with a Penn PCP, we will use a default centralized referral model to engage PCPs to sign a referral for their patients to see a lipid specialist. Arm 2) Direct to Patient: For patients without a PCP at Penn, we will conduct direct outreach to the patients to invite them to schedule a free telehealth appointment with a lipid specialist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without a primary care physician within the UPHS health system (Experimental): Patients without a primary care physician within the UPHS health system will receive direct outreach from the study team to invite them to schedule a visit with a lipid specialist for a formal evaluation of FH.
  Interventions: Behavioral: Inviting patients to complete a telehealth appointment with a lipid specialist for an FH evaluation
- Patients with a primary care physician within the UPHS health system (Experimental): For patients with a primary care physician within the UPHS health system, their primary care physicians will be asked to review and sign physician referrals to a lipid specialist and invite patients to schedule a visit with a lipid specialist for a formal evaluation of FH.
  Interventions: Behavioral: Testing centralized referral mechanism for PCPs; Behavioral: Inviting patients to complete a telehealth appointment with a lipid specialist for an FH evaluation

INTERVENTIONS:
Behavioral: Testing centralized referral mechanism for PCPs — For patients with a Penn PCP, we are testing a centralized referral mechanism to increase the number of referrals to preventive cardiology (default/opt out referrals)
  For default/opt out: PCPs will receive a pended order for a referral for their patient to see a lipid specialist for a formal FH evaluation. Not interacting with the pended order or accepting the pended order will indicate that the referral to a lipid specialist should be placed.
  Arms: Patients with a primary care physician within the UPHS health system
Behavioral: Inviting patients to complete a telehealth appointment with a lipid specialist for an FH evaluation — All eligible patients will be informed that they have been identified by the FIND FH tool as potentially having familial hypercholesterolemia. All patients will be invited to schedule a telehealth appointment with a lipid specialist for a formal evaluation for FH.

SUMMARY:
The goal of this study is to identify individuals at high risk of FH, and to encourage the appropriate diagnosis and treatment of individuals at high risk of FH through the use of implementation science and behavioral economics principles.

Phase 1: Applying the FIND FH tool to the health system EHR and gathering data for pilot development; Phase 2: Pilot development and implementation; Phase 3: Conduct a large-scale pragmatic trial consistent with recommendations and learnings from the pilots in Phase 2

DETAILED DESCRIPTION:
Phase 1:

Aim 1: Adjusting and refining the application of the FIND FH tool to the UPHS EHR database Aim 2: Identifying the barriers and facilitators to making a diagnosis of FH and initiating or intensifying therapy for individuals with FH through qualitative interviews with clinicians and patients and creating a behavioral roadmap to inform the implementation approaches to test in the pilots

Phase 2:

Aim 1: Co-design implementation strategies using behavioral economics in partnership with the Family Heart Foundation Aim 2: Pilot implementation strategies with an enrollment goal of 80 patients total (40 per pilot) who have been flagged by the FIND FH tool as having probable FH to ascertain feasibility, acceptability, and appropriateness

Phase 3: Conduct a large-scale pragmatic trial consistent with recommendations and learnings from the pilots in Phase 2

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient at Penn Medicine
* Must have been flagged by the FIND FH tool as having a high probability of FH
* First language is English
* Resides in PA or NJ

Exclusion Criteria:

* Already have been clinically diagnosed with FH using the proper ICD-10 code
* Currently see a lipid specialist at Penn Medicine
* Pass study clinician's Study Validity Check

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of flagged patients diagnosed with FH (familial hypercholesterolemia) as a result of the intervention | Day 1 - post intervention study visit
  Patients will be evaluated for familial hypercholesterolemia (FH), an underdiagnosed genetic type of high cholesterol. An FH diagnosis will be defined using the Dutch Lipid Clinic Network Diagnostic (DLCN) Criteria for FH (Unlikely, Possible, Probable, Definite). The clinician will also make a clinical assessment of FH informed by the DLCN score and clinical expertise from the appointment.

SECONDARY OUTCOMES:
Proportion of patients that have a change to their lipid management because of the intervention | Day 1 - post intervention study visit
  Defined as the proportion of patients that start (or are prescribed) statins, ezetimibe, PCSK9 inhibitors, or have any intensification of any lipid lowering medications as a result of the visit with the lipid specialist for patients that qualify at the time of the appointment with the lipid specialist.
Proportion of patients that have a change to their lipid management among patients that were candidates for a change to their lipid management because of the intervention | Day 1 - post intervention study visit
  Defined as the proportion of patients that start (or are prescribed) statins, ezetimibe, PCSK9 inhibitors, or have any intensification of any lipid lowering medications as a result of the visit with the lipid specialist for patients that qualified and were not already optimally treated at the time of the appointment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No